CLINICAL TRIAL: NCT05963074
Title: Multicohort Study to Customize Ibrutinib Treatment Regimens for Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study to Customize Ibrutinib Treatment Regimens for Participants With Previously Untreated Chronic Lymphocytic Leukemia
Acronym: TAILOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 54179060CLL2032; 54179060CLL2032 (Other: Janssen Research & Development, LLC); 2023-504044-34-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1a: Ibrutinib Lead-in+Fixed Duration Ibrutinib+Venetoclax (Experimental): Participants will receive ibrutinib 420 milligrams (mg) capsule every day (QD) for a lead-in of 3 cycles (1 cycle = 28 days). From Cycle 4, venetoclax 400 mg tablet dose ramp-up (from 20 to 400 mg over 5 weeks) will begin, and venetoclax 400 mg QD will be administered with ibrutinib 420 mg QD, orally for 12 cycles through Cycle 15.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Cohort 1b: Ibrutinib Lead-in+Fixed Duration Ibrutinib+Venetoclax (Experimental): Participants will receive ibrutinib 420 mg capsule QD for a lead-in of 3 cycles (1 cycle = 28 days). From Cycle 4, venetoclax 400 mg tablet dose ramp-up (from 20 to 400 mg over 5 weeks) will begin and ibrutinib dose will be reduced to 280 mg and will be administered QD, venetoclax 400 mg tablets QD will be administered with ibrutinib 280 mg for 12 cycles through Cycle 15.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Cohort 2a: Continuous Ibrutinib Monotherapy (Experimental): Participants will receive ibrutinib 420 mg QD (or last tolerated dose) until disease progression (PD) or unacceptable toxicity.
  Interventions: Drug: Ibrutinib
- Cohort 2b: Continuous Ibrutinib Monotherapy (Experimental): Participants will receive ibrutinib 420 mg QD for 1 cycle (1 cycle = 28 days) followed by Ibrutinib 280 mg QD (or last tolerated dose) and continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib capsules will be administered orally.
  Other Names: JNJ-54179060, IMBRUVICA
Drug: Venetoclax — Venetoclax tablets will be administered orally.
  Other Names: VENCLEXTA, VENCLYXTO
  Arms: Cohort 1a: Ibrutinib Lead-in+Fixed Duration Ibrutinib+Venetoclax; Cohort 1b: Ibrutinib Lead-in+Fixed Duration Ibrutinib+Venetoclax

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ibrutinib + venetoclax (I+V) and ibrutinib monotherapy regimens in which dosing of ibrutinib is either proactively reduced or reactively modified in response to adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia/ small lymphocytic lymphoma (CLL/SLL) as per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 diagnostic criteria
* For ibruinib + venetocIax (I+V) cohorts: eastern cooperative oncology group (ECOG) performance status of 0-1. For ibrutinib monotherapy cohorts: ECOG performance status of 0-2
* Measurable nodal disease by computed tomography (CT), defined as at least 1 lymph node greater than and equal to (>=) 1.5 centimeters (cm) in longest diameter
* A participant using oral contraceptives must use an additional contraceptive method
* A participant must agree not to be pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or until 1 month after last dose or per local label if more conservative (for example, 3 months in European Union or Canada and 1 month in United States)

Exclusion Criteria:

* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura, such as those participants with a declining hemoglobin level or platelet count secondary to autoimmune destruction within the 4 weeks prior to first dose of study treatment, or the need for prednisone greater than (>) 20 milligrams (mg) daily (or corticosteroid equivalent) to treat or control the autoimmune disease
* Known bleeding disorders (example, von Willebrand's disease or hemophilia)
* Stroke or intracranial hemorrhage within 6 months prior to enrollment
* Known or suspected Richter's transformation or central nervous system (CNS) involvement
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class II, III, or IV congestive heart failure as defined by the New York Heart Association Functional Classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-03-19 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (ORR) | Up to 5 years
  Best ORR is defined as the percentage of participants who achieve complete remission (CR), complete remission with an incomplete marrow recovery (CRi), nodular partial remission (nPR), or partial remission (PR) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria as assessed by investigator.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | Up to 5 years
  CR rate is defined as the percentage of participants achieving a best overall response of CR or CRi per iwCLL 2018 criteria as assessed by investigator.
Duration of Response (DOR) | Up to 5 years
  DOR is defined as the duration in days from the date of initial documentation of PR or better to the date of first documented evidence of PD or death.
Progression Free Survival (PFS) | Up to 5 years
  PFS by investigator assessment is defined as the duration from date of randomization to date of PD or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from date of randomization to date of death from any cause.
Cohorts 1a and 1b: Minimal Residual Disease (MRD) Negative Rate | Up to 5 years
  MRD-negative rate is defined as the percentage of participants who reach MRD-negative status (that is, less than [<] 1 chronic lymphocytic leukemia (CLL) cell per 10,000 leukocytes or <0.01 percentage [%]) in the peripheral blood.
Number of Participants with Adverse Events (AEs) | Up to 5 years
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 5 years
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Percentage of Participants with Rate of Discontinuation due to AEs | Up to 5 years
  Percentage of participants with rate of discontinuation due to AEs will be reported.
Percentage of Participants with Dose Reduction due AEs | Up to 5 years
  Percentage of participants with dose reduction due AEs will be reported.
Adherence Rates | Up to 5 years
  The adherence rate is defined as the percentage of total dose taken over the total dose prescribed.
Duration of Treatment | Up to 5 years
  Duration of treatment is defined as the time period in days between the date of first study treatment administration and date of last administration.
Time to Worsening as Measured by EuroQol 5 Dimension 5 Level Questionnaire (EQ-5D-5L) | Up to 5 years
  Time to worsening is defined as time interval (months) from randomization to first observation of deterioration. Time to worsening as measured by EQ-5D-5L will be reported.
Time to Worsening as Measured by European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC QLQ)-C30) | Up to 5 years
  Time to worsening is defined as time interval from randomization to first observation of deterioration. Time to worsening as measured by EORTC QLQ-C30 will be reported.
Time to Worsening as Measured by EORTC QLQ-CLL17 | Up to 5 years
  Time to worsening is defined as time interval from randomization to first observation of deterioration. Time to worsening as measured by EORTC QLQ-CLL17 will be reported.
Time to Worsening as Measured by Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Total Score | Up to 5 years
  Time to Worsening is defined as time interval (months) from randomization to first observation of deterioration. Time to worsening as measured by FACIT-fatigue total score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (74):
- United States (32):
  - The Oncology Institute Clinical Research, Cerritos, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - SLO Oncology and Hematology Health Center, San Luis Obispo, California
  - Providence Medical Foundation, Santa Rosa, California
  - PIH Health Hospital, Whittier, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Mount Sinai Medical Center Campus, Miami Beach, Florida
  - The Oncology Institute, North Miami Beach, Florida
  - Mid Florida Hematology Oncology, Orange, Florida
  - Boise VA Medical Center, Boise, Idaho
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Iowa City VA Health Care System, Iowa City, Iowa
  - Minnesota Oncology Hematology P A, Minneapolis, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Renovatio Clinical, El Paso, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Texas Oncology-Gulf Coast, The Woodlands, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Virginia Cancer Specialists, Manassas, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - VA Puget Sound Healthcare System, Seattle, Washington
  - Northwest Cancer Specialists PC, Vancouver, Washington
- Canada (2):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Niagara Health System, St. Catharines, Ontario
- Czechia (6):
  - Fakultni nemocnice Brno, Brno-Bohunice
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Ustav Hematologie A Krevni Transfuze, Prague
- France (6):
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Nantes, Nantes
  - Hopital Pitie Salpetriere, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Reims, Reims
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Gyor Moson Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Szabolcs Szatmar Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - University of Szeged, Szeged
- Italy (11):
  - U.O. Ematologia Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliero-Universitaria di Ferrara Arcispedale Sant Anna, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Maggiore della Carita, Novara
  - Universita degli Studi di Padova Azienda Ospedaliera di Pa, Padua
  - Ospedale Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliera di Perugia Ospedale S.Maria della Misericordia, Perugia
  - Ematologia Fondazione Univ. Policlinico Gemelli Università Cattolica del Sacro Cuore, Roma
  - Umberto I Policlinico di Roma, Roma
- Poland (7):
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli, Lublin
- Spain (6):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency